CLINICAL TRIAL: NCT05805644
Title: Effects of Robot-mediated Impairment-Oriented and Task-Specific Training on Upper Limb Outcomes Post Stroke (RMT-Stroke Outcomes)
Brief Title: Robot Mediated Therapy-Upper Limb Outcomes in Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChangiGH1
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Care Provider, Outcomes Assessor
Masking Description: To prevent subversion of the allocation sequence, study team members who enroll patients to the trial will be distinct and kept separate from the study team member that perform the randomization. We will establish the procedures to maintain separation between study team members that assess the outcomes, and those that perform group assignment. At the start of every assignment, patients will be reminded to not reveal their treatment assignment by referring to elements of the treatment that are unique to their treatment group.
  Functional outcome scales are performed by blinded therapists who work in the unit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot mediated Impairment-oriented training(RMIT) (Experimental): Participant receives 20 hours of robot mediated impairment-oriented training applied via the Optimo Regen
  Interventions: Device: Robot mediated upper limb therapy
- Robot mediated impairment-oriented and task-specific training (RMIT+RMTT) (Experimental): Participant receives a total of 20 hours of robotic therapy. 10 hours will be in the form of RMIT and 10 hours in the form of RMTT
  Interventions: Device: Robot mediated upper limb therapy

INTERVENTIONS:
Device: Robot mediated upper limb therapy — The OR is classified as a Class A device with the Health Sciences Authority. The OR is capable of delivering RMIT as well as RMTT. It can provide zero, partial or full assistance to the patient to complete the movement or task. Its teach-and-follow mode allows a movement to be performed by the therapist, with the device then "replaying" the movement at either zero, partial or full assistance for the patient.
  Impairment oriented training will focus on the following movements:
  1. Diagonal movement
  2. Shoulder abduction
  3. Shoulder adduction
  4. Shoulder flexion
  5. Shoulder extension
  6. Elbow flexion
  7. Elbow extension
  Task-specific training will focus on the following activities:
  1. Picking up a cup/glass by the side and drink
  2. Brushing hair
  3. Cleaning unaffected upper limb (hand to arm)
  4. Wiping table
  5. Wiping wall
  6. Sliding card on table to a designated location
  7. Clipping a clothe peg

SUMMARY:
This study aims to determine the clinical outcomes of stroke patients who are provided with adjunctive robot-mediated task specific therapy(RMTT) and robot-mediated impairment training (RMIT) as compared to those who are provided with adjunctive RMIT.

DETAILED DESCRIPTION:
Stroke is among the top 10 causes of hospitalisation in Singapore1. Approximately 630 stroke patients were transferred to our inpatient rehabilitation unit in 2021. Upper limb impairments are common after stroke2 and may result in loss of function, including self-care activities. Intensity of therapy is thus important for post-stroke recovery. A Cochrane overview of systematic reviews suggested that arm function can be improved by providing at least 20 hours of additional repetitive task training to patients3. However, providing sufficient therapy remains a challenge due to various reasons4, including manpower shortages. Robotic-mediated rehabilitation is an innovative exercise-based therapy using robotic devices that enables the implementation of highly repetitive, intensive, adaptive, and quantifiable physical training.

The RATULS trial5 showed that neither robot-assisted training using the MIT-Manus robotic gym nor an enhanced upper limb therapy (EULT) programme based on repetitive functional task practice improved upper limb function after stroke, as compared to usual care, for patients with moderate-to-severe upper limb functional limitations. It was suggested that further research was needed to find ways to translate the improvements in upper limb impairments seen with robot-assisted therapy into upper limb function and their activities of daily living (ADLs).

In a systematic review and meta-analysis on the effects of robot-assisted therapy on the upper limb, it was found that although there were improvements in strength, this was not translated to improvements in activities of daily living6. Additional transition to task training (facilitated by therapists) had been added to robot-mediated impairment training (RMIT) in various studies7,8. In a study by Hung8, robot-assisted therapy combined with occupational therapist (OT)-facilitated task specific training was found to be superior to robot-assisted therapy combined with OT-facilitated impairment-oriented training. Task-specific training consists of repetitively practising the tasks that are most relevant to the patient and their personal context, whereas impairment-oriented therapy emphasises remediation of motor deficits with a focus on single joint movements at a time.

A study that investigated Reharob, a robotic device used to assist patients living with chronic stroke in performing 5 ADLs, showed that patients had significant improvements on the Fugl-Meyer Assessment - Upper Extremity (FMA-UE), Action Research Arm Test (ARAT) and Functional Independence Measure (FIM)9. This is the only study that has been found addressing robot-mediated task-specific training thus far (RMTT).

This study aims to determine the clinical outcomes of stroke patients who are provided with both RMTT and robot-mediated impairment training (RMIT) in addition to conventional therapy, as compared to those who are provided with only adjunctive RMIT. From a review of the prevalent literature, there has been no study on the comparison of RMTT + RMIT against RMIT alone. A search for RMTT only yielded the study on Reharob, but the robot only administered RMTT and not RMIT.

The target patients would be those with acute stroke undergoing rehabilitation in an acute inpatient rehabilitation unit. Robotic therapy can continue when they are discharged, in the outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of stroke as evidenced by CT/MRI findings
2. First-ever stroke (ischaemic or haemorrhagic)
3. Upper limb weakness and an FMA-UE score of 16-53 (severe to moderate: 16-34. moderate to mild: 35-53)12,13
4. Cognitively intact to follow instructions
5. Medically stable to participate
6. Consent given
7. Age 21 and above

Exclusion Criteria:

1. Fractures or other musculoskeletal issues that render the use of the robotic device unsuitable 2. Involvement in another concurrent upper limb study 3. Wounds that do not allow donning of the device 4. Severe spasticity 5. Cognitive impairment (MMSE ≤20) 6. Inability to follow instructions 7. Severe osteoporosis 8. Infectious diseases that require the patient to be isolated in a single room eg airborne diseases

-

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of FMA-UE(Fugl Meyer Assessment for Upper Extremity) from baseline | baseline, 1 month and 3 months post commencement of intervention
  30 items assessing motor function and 3 items assessing reflex function (0-66, higher scores indicates better outcomes)

SECONDARY OUTCOMES:
Change of FMA-UA( Fugl Meyer Assessment-Upper Arm) from baseline | baseline, 1 month and 3 months post commencement of intervention
  subset of FMA-UE( 0-36, higher score indicates better outcomes)
Change of FMA-W/H (Fugl Meyer Assessment- Wrist/Hand) from baseline | baseline, 1 month and 3 months post commencement of intervention
  subset of FMA-UE (0-30, higher scores indicates better outcomes)
Change of FAT( Frenchay Arm Test) from baseline | baseline, 1 month and 3 months post baseline
  Upper limb functional assessment (0-5, higher score indicates better outcomes)
Change of FIM (Functional Independence Measure) from baseline | baseline, 1 month, 3 months post baseline
  Functional outcome measure, mainly used in inpatient setting (18-126, higher score indicates better outcomes)
Change of MMT( manual muscle testing) from baseline | baseline, 1 month and 3 months post baseline
  Using the Medical Research Council scale (0-5, higher indicates better outcomes)
Change of MAS (Modified Ashworth Scale) from baseline | baseline, 1 month and 3 months post baseline
  spasticity assessment scale (0-4, lower indicates better outcomes)
Change of EQ5D from baseline | baseline, 1 month and 3 months post baseline
  Quality of Life Questionaire (0-100, higher score indicates better outcomes)
Change of HADS (Hospital Anxiety and Depression Scale) from baseline | baseline, 1 month and 3 months post baseline
  Masurement of mood (0-42, more than 8 points in each subcategory indicates considerable symptoms of anxiety or depression)
Change of patient satisfaction survey from baseline | baseline, 1 month and 3 months post baseline
  Patient satisfaction survey (8-40), higher score denotes good outcome)
Difference in the presence of adverse effects | baseline, 1 month and 3 months post baseline
  fatigue, pain, injuries (present or absent. Absent denotes better outcome)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Conroy SS, Wittenberg GF, Krebs HI, Zhan M, Bever CT, Whitall J. Robot-Assisted Arm Training in Chronic Stroke: Addition of Transition-to-Task Practice. Neurorehabil Neural Repair. 2019 Sep;33(9):751-761. doi: 10.1177/1545968319862558. Epub 2019 Jul 22. PMID 31328671
- [Result] Mehrholz J, Pohl M, Platz T, Kugler J, Elsner B. Electromechanical and robot-assisted arm training for improving activities of daily living, arm function, and arm muscle strength after stroke. Cochrane Database Syst Rev. 2018 Sep 3;9(9):CD006876. doi: 10.1002/14651858.CD006876.pub5. PMID 30175845
- [Result] Hung CS, Hsieh YW, Wu CY, Lin KC, Lin JC, Yeh LM, Yin HP. Comparative Assessment of Two Robot-Assisted Therapies for the Upper Extremity in People With Chronic Stroke. Am J Occup Ther. 2019 Jan/Feb;73(1):7301205010p1-7301205010p9. doi: 10.5014/ajot.2019.022368. PMID 30839256